CLINICAL TRIAL: NCT00242307
Title: A Confirmatory Study of APTA-2217 in Adult Patients With Bronchial Asthma (A Placebo-controlled Double-blind Comparative Study)
Brief Title: Efficacy and Safety of Roflumilast in Japanese Patients With Bronchial Asthma (20 to 70 y) (APTA-2217-05)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APTA-2217-05
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-09

CONDITIONS: Bronchial Asthma
Keywords: Asthma; Roflumilast; phosphodiesterase 4 inhibitor
MeSH Terms: conditions — Asthma | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
The aim of the study is to investigate the effect of roflumilast (APTA-2217) on lung function in patients with asthma. Roflumilast will be administered orally once daily. The study duration consists of a baseline period (2 to 4 weeks) and a treatment period (24 weeks). The study will provide further data on safety, tolerability, and effectiveness of roflumilast.

ELIGIBILITY:
Main inclusion criteria:

* Adult patients with bronchial asthma meeting the Guideline for Prevention and Control of Asthma 2003 (JGL 1998, revised 2nd edition)
* No change in asthma treatment during the last 4 weeks prior to the registration
* Non-smokers or ex-smokers for 12 months or more
* %FEV1 ranging between 60 and 80%

Main exclusion criteria:

* Patients with poorly controlled asthma
* Inhalation therapy exceeding low dose during 4 weeks prior to the registration
* Concurrent respiratory diseases such as COPD considered to affect the efficacy evaluation

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2004-05; Primary Completion 2006-09 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
change in lung function parameters.

SECONDARY OUTCOMES:
pulmonary function test (spirometry), asthma symptoms, rescue medication, evaluation of QOL, asthma exacerbation, adverse events, pharmacokinetics.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Nycomed Japan and Mitsubishi Tanabe Pharma Corporation, Osaka, Japan

REFERENCES:
- See also: APTA-2217-05-RDS-2008-12-17.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4454&filename=APTA-2217-05-RDS-2008-12-17.pdf